CLINICAL TRIAL: NCT05255588
Title: A Multicenter, Single-blind, Prospective Clinical Trial to Evaluate the Clinical Performance of EarlyTect® CRC Test for the Early Detection of Colorectal Cancer in the Stool DNA From High-risk Group
Brief Title: A Stool DNA-based SDC2 Methylation Test for the Early Detection of Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Genomictree, Inc. (Industry)
Collaborators: Soon Chun Hyang University (Other); Gangnam Severance Hospital (Other); Kyung Hee University Hospital at Gangdong (Other); Kangbuk Samsung Hospital (Other); Kyung Hee University Hospital (Other); Keimyung University Dongsan Medical Center (Other); Korea University Anam Hospital (Other); Pusan National University Hospital (Other); The Catholic Univ. of Korea Bucheon ST. Mary's Hospital (Unknown); Samsung Medical Center (Other); Seoul National University Hospital (Other); Asan Medical Center (Other); Wonju Severance Christian Hospital (Other); Severance Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NEXT-CRC
Record Dates: First submitted 2022-02-16; First posted 2022-02-24 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer; Advanced Colorectal Neoplasm; Advanced Adenomas; Non-neoplastic Polyps; Non-advanced Adenomas
Keywords: Colorectal cancer; SDC2; Methylation biomarker; EarlyTect® CRC test; Stool
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual stool samples may be archived for further research. Clinical data and samples will be kept in a manner that preserves anonymity of the subjects, using the subject ID as the only tracking information. Specimens will be stored at Genomictree and may be used for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort: Subjects who are at high-risk (Asia Pacific Colorectal Screening Score ≥4.0) of developing CRC aged ≥40
  Interventions: Device: EarlyTect® CRC test

INTERVENTIONS:
Device: EarlyTect® CRC test — A highly accurate and sensitive real time PCR employing Linear Target Enrichment and Quantitative Methylation-Specific PCR (LTE/qMSP) for measuring SDC2 methylation in stool DNA to detect CRC.

SUMMARY:
The primary objective of this clinical trial is to determine the sensitivity and specificity of the EarlyTect® CRC test for detecting CRC, using colonoscopy as the reference method.

The secondary objective is to compare the clinical performance of EarlyTect® CRC test with a commercially available Fecal Immunochemical Test (FIT), with respect to CRC. By histopathological examination, lesions identified during colonoscopy will be confirmed as malignant or precancerous by histological examination.

DETAILED DESCRIPTION:
A multicenter, single-blind, prospective clinical trial is being conducted to evaluate the clinical performance of EarlyTect® CRC test. Subjects who are at high-risk (Asia Pacific Colorectal Screening Score ≥4.0) of developing CRC who are eligible for inclusion criteria will be asked to collect a stool sample and EarlyTect® CRC and FIT tests will be performed. For confirmation of the diagnosis and tumor staging, representative histopathology slides obtained from curative surgery and representative histopathology slides from tissue biopsied or excised during colonoscopy may be retrieved and examined by the central pathology laboratory. Methylation status of SDC2 in stool DNA is measured by a highly accurate and sensitive real time PCR that employs Linear Target Enrichment (LTE) and quantitative Methylation-Specific PCR (qMSP)(LTE-qMSP).

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled into the study must meet the following criteria:

* Individuals who agree to voluntarily sign an informed consent prior to the initiation of screening
* Adults aged ≥ 40 years
* Subjects who are at high-risk (Asia Pacific Colorectal Screening (APCS) Score: 4.0~7.0) of developing CRC
* Subjects who are able and willing to undergo colonoscopy screening within 12 months of consent among individuals who reserved a visit in the division of gastroenterology or health check-up.

Exclusion Criteria:

Subjects will be excluded from enrolling into the study if any of the following criteria are met:

* Individuals who do not agree to voluntarily sign an informed consent prior to the initiation of screening
* Adults aged < 40 years
* Subjects who are not at high-risk (APCS Score ≤ 3.0) of developing CRC
* Subjects who will not undergo colonoscopy screening within 12 months of consent
* Subjects who have had a positive FIT or fecal occult blood test within the previous 2 weeks
* Colorectal cancer patients who did not underwent curative treatment
* Subjects who have had a prior history of colorectal resection
* Subjects who have had overt rectal bleeding or melena within the previous 2 weeks
* Subjects who have a family history or a prior history of hereditary CRC or colorectal neoplasm: Lynch syndrome (HNPCC), familial adenomatous polyposis, MUTYH-associated polyposis, Juvenile polyposis syndrome, Peutz-Jeghers syndrome, and serrated polyposis syndrome, etc.
* Subjects who have inflammatory bowel diseases including Crohn's disease, ulcerative colitis or Behcet disease
* Subjects who participated in any "interventional" clinical study within the previous 30 days
* Subject has any condition which, in the opinion of the medical staff should preclude participation in the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are at high-risk (Asia Pacific Colorectal Screening Score ≥4.0) of developing CRC
Sampling Method: Non-Probability Sample
Enrollment: 2358 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the EarlyTect® CRC test for detecting CRC compared to the colonoscopy, both in terms of detecting CRC. | 18 months
  The reference method is the colonoscopy, and lesions will be assessed histopathologically.
  EarlyTect® CRC test includes a measurement of SDC2 methylation and COL2A1 as a DNA control. SDC2 methylation in stool DNA will be assessed quantitatively by LTE/qMSP. The results will be dichotomized by the CT (cycle threshold) cutoff value as either positive or negative. Sensitivity = 100*(positive SDC2 methylation test/positive colonoscopy), Specificity = 100*(negative SDC2 methylation test/negative colonoscopy).

SECONDARY OUTCOMES:
Sensitivity of EarlyTect® CRC for detecting advanced colorectal adenoma (Adenomas ≥1.0 cm, villous adenomas or high-grade dysplasia) | 18 months
  Sensitivity for detecting adenomas ≥1.0 cm
  * Sensitivity of EarlyTect® CRC for detecting villous adenomas
  * Sensitivity of EarlyTect® CRC for detecting high-grade dysplasia
Sensitivity of EarlyTect® CRC for detecting advanced colorectal neoplasm | 18 months
  Sensitivity for detecting adenomas ≥1.0 cm
Sensitivity of EarlyTect® CRC for detecting non-advanced adenomas | 18 months
  Sensitivity for detecting non-adenomas <1.0 cm
Sensitivity and specificity of combined FIT and EarlyTect® CRC tests in detecting CRC | 18 months
  Sensitivity and specificity of combined FIT and EarlyTect® CRC tests in detecting CRC
Sensitivity of EarlyTect® CRC for detecting advanced colorectal serrated lesions | 18 months
  Sensitivity of EarlyTect® CRC for detecting advanced colorectal serrated lesions
Clinical specificity of EarlyTect® CRC when patients with non-advanced adenomas and non-advanced colorectal serrated lesions are included in control group | 18 months
  Clinical specificity of EarlyTect® CRC when patients with non-advanced adenomas and non-advanced colorectal serrated lesions are included in control group
Clinical sensitivity of the EarlyTect® CRC for detecting Tis | 18 months
  Clinical sensitivity of the EarlyTect® CRC for detecting colorectal cancer with Tis

CONTACTS AND LOCATIONS:
Locations (1):
- Soon Chun Hyang University Hospital Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oh TJ, Oh HI, Seo YY, Jeong D, Kim C, Kang HW, Han YD, Chung HC, Kim NK, An S. Feasibility of quantifying SDC2 methylation in stool DNA for early detection of colorectal cancer. Clin Epigenetics. 2017 Dec 4;9:126. doi: 10.1186/s13148-017-0426-3. eCollection 2017. PMID 29225717
- [Background] Han YD, Oh TJ, Chung TH, Jang HW, Kim YN, An S, Kim NK. Early detection of colorectal cancer based on presence of methylated syndecan-2 (SDC2) in stool DNA. Clin Epigenetics. 2019 Mar 15;11(1):51. doi: 10.1186/s13148-019-0642-0. PMID 30876480